CLINICAL TRIAL: NCT01613365
Title: Oropharyngeal and Nasopharyngeal Decontamination With Chlorhexidine Gluconate in the Reduction of the Postoperative Morbidity and Mortality After Major Pulmonary Resections: a Multicentric, Prospective, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Oropharyngeal and Nasopharyngeal Decontamination With Chlorhexidine Gluconate in the Reduction of the Postoperative Morbidity and Mortality After Major Pulmonary Resections
Acronym: CHLORHEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-004536-63; 2011-24 (Other: AP HM)
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Infections and Respiratory Infectious
MeSH Terms: conditions — Infections | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- chlorhexidine gluconate (Experimental)
  Interventions: Drug: Chlorhexidine Gluconate
- placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — Oropharyngeal and nasopharyngeal decontamination with Chlorhexidine Gluconate
  Arms: chlorhexidine gluconate
Drug: Placebo — Oropharyngeal and nasopharyngeal decontamination with placebo
  Arms: placebo

SUMMARY:
Despite improvement of per and postoperative management, major pulmonary surgery continues to carry out a high morbidity with a significant mortality. Among postoperative complications, respiratory failures (nosocomial pneumonia, ARDS) are currently the most frequent and serious, as well as being the primary cause of hospital death, after major pulmonary resections. Vast majority of these complications are notoriously infectious and should be considered as hospital-acquired infections. These complications result in a dramatic increased of substantial hospital costs in term of length of hospital stay, antibiotics and morbidity. Current management of these complications stands on antibiotics, oxygen supply and physiotherapy. In severe case, a ventilatory support (invasive or non invasive) is justify in near 25 % of cases.

Recent data have suggested that proximal airways colonizations could be an essential first step in the pathogenesis of theses respiratory failures. Previous works have long demonstrated that bacterial colonization was frequent between 21 to 40 % in lung cancer patients. These colonizations could act as a major predisposing factor to these postoperative respiratory failures. Because distal airways and lung parenchyma are free from bacteria at the moment of the surgery, respiratory complications should be the result from contamination by potential microorganisms belonging the upper aero-digestive tract. Consequently, decontamination of the oropharyngeal and nasopharyngeal cavities before and during the first days after surgery could have a beneficial advantage in the prevention of these complications. This decontamination has been demonstrated to be effective in critically-ill patients in intensive care unit, in cardiac surgery and in esophageal surgery. Decontamination of oropharynx and nasopharynx with Chlorhexidine Gluconate has significantly reduced the rate of postoperative global hospital-acquired infections and respiratory infectious as well. To date, data on the efficacy of this decontamination protocol in major pulmonary resections are not available.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women over 18 years
* Submitted to major pulmonary resections for primary lung cancer or pulmonary metastasis
* Anatomical resections (segmentectomy, lobectomy, pneumonectomy)
* With mediastinal lymph node dissection.
* Patient fit for operation
* After informed consent

Non inclusion criteria:

* Patients < 18 years
* Pulmonary infectious lesions
* Recent respiratory infections
* Tracheostomy
* Swallow difficulties
* Need for non-invasive ventilation before surgery
* Documented sensibility to Chlorhexidine
* Previous ENT cancer
* Previous thoracic surgery
* Patients with an oral assessment score (OAG) >9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
proportion of patients requiring ventilatory support | 36 MONTHS

SECONDARY OUTCOMES:
occurrence of documented hospital-acquired respiratory infections | 36 MONTHS
occurrence of documented non-respiratory hospital-acquired infections | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille; D'JOURNO BENOIT, Principal Investigator — AP HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] D'Journo XB, Falcoz PE, Alifano M, Le Rochais JP, D'Annoville T, Massard G, Regnard JF, Icard P, Marty-Ane C, Trousse D, Doddoli C, Orsini B, Edouard S, Million M, Lesavre N, Loundou A, Baumstarck K, Peyron F, Honore S, Dizier S, Charvet A, Leone M, Raoult D, Papazian L, Thomas PA. Oropharyngeal and nasopharyngeal decontamination with chlorhexidine gluconate in lung cancer surgery: a randomized clinical trial. Intensive Care Med. 2018 May;44(5):578-587. doi: 10.1007/s00134-018-5156-2. Epub 2018 Apr 18. PMID 29671041